CLINICAL TRIAL: NCT03736876
Title: About Us: A Healthy Relationships Program for Vulnerable Youth
Brief Title: A Healthy Relationships Program for Vulnerable Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Collaborators: Family and Youth Services Bureau (Unknown); San Diego State University (Other); California School-Based Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90 AP2682-01-00
Record Dates: First submitted 2018-08-22; First posted 2018-11-09 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy, Unplanned; Sexually Transmitted Diseases
Keywords: Youth; Adolescents; Teens; Healthy Relationships; Unintended Pregnancy; Teen Pregnancy; Sexually Transmitted Infections; Sexually Transmitted Diseases; Sexual Health Education; School-Based Health Center; Randomized Controlled Trial
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Multi-site independent randomized group treatment trial (IGRT). 1,209 youth randomized to intervention or control conditions within schools. Sample accrues over 2.5 years (Years 2-4)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): These students will receive About Us, an innovative, healthy relationship intervention. The program includes 10 lessons that blend group-based activities with online activities implemented in school-based health centers.
  Interventions: Behavioral: About Us
- Delayed intervention (control group) (No Intervention): These students will receive the business-as--usual condition (e.g., the standard health education that is provided by the school during the study period), and will receive the intervention once the study period has concluded.

INTERVENTIONS:
Behavioral: About Us — Each program session includes an initial soap opera-like story to build interest and illustrate key concepts, 2-3 group-based activities with reflection, individual app-based work on tablets to allow for personalization of the content, and a group-based debrief to reflect on the day and reinforce key messages. The group-based content is delivered by trained facilitators from the participating school-based health centers. The app-based content is housed on a secure website and accessed through tablets with unique log-ins for each participant. Activities are completed individually during the session (e.g., completing a poll; watching and responding to a brief video). Several lessons include homework activities that encourage communication between students and a caring adult.
  Arms: Treatment group

SUMMARY:
Developed from a piloted intervention and based on scientific evidence, About Us is an innovative healthy relationships intervention that promotes positive adolescent romantic relationships and use of condoms and highly effective contraceptives if having sex. The program includes 10 lessons (2 that are between 30-45 minutes long 8 that are 50 minutes long) that blend group-based activities with online activities implemented in a small group format with students in grades 9 or 10 who have parental consent and provide assent to take part. The program will be implemented in school-based health centers (SBHCs).

Primary research question:

1. Nine months following the end of the program, what is the impact of About Us relative to the standard of care on:

   1.1. Rates of vaginal or anal sex without condoms in the past three months?

   Secondary research questions:
2. Three and nine months following the end of the program, what is the impact of About Us relative to the standard of care on:

   2.1. Rates of abstinence from vaginal or anal sex in the past three months? 2.2. Frequency of communicating without abuse? 2.3. Utilization of school-based health center services? 2.4. Rates of behavioral willingness and attitudes toward birth control?

   Exploratory research questions:
3. Three and nine months following the end of the program, what is the impact of About Us relative to the standard of care on:

   3.1. The psychosocial variables stemming from the theoretical framework (e.g., attitudes toward condom and contraceptive use, normative beliefs, perceived self-efficacy to use condoms or have difficult conversations) and enumerated in the logic model.

   3.2. Outcomes listed above within key sub-groups including those defined by sex (male/female), race/ethnicity, and exposure to violence;
4. Among those receiving About Us, how do effect sizes for the primary and secondary behavioral outcomes vary by dosage?

DETAILED DESCRIPTION:
Students will be screened for eligibility through each school-based health center (SBHC) by SBHC staff, and those participants meeting the screening eligibility requirements (previous exposure to violence and/or previous or current involvement in a romantic relationship) will be offered a parental consent form and informational packet. Consent forms will be available in English and Spanish. Pending parental consent and youth assent, students will be randomized into either the intervention or control group.

ELIGIBILITY:
Inclusion Criteria:

* The target population includes 9th or 10th grade students from participating schools who meet at least one of the following inclusion criteria based on their responses to a school-wide health assessment:

  1. prior exposure to violence;
  2. prior or current experience with a romantic relationship.

Any student answering "yes" to either criteria would be eligible to take part in the study. Only those who have parent consent and assent would be enrolled.

Exclusion Criteria:

* Those students without parental consent;
* If siblings are eligible to participate, the sibling who returns the signed consent form first will be admitted into the study. Any other eligible siblings will be excluded.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 550 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Rates of vaginal or anal sex without condoms | 9 months post intervention
  Reported number of times having had vaginal or anal sex without using condoms or insertive condoms.

SECONDARY OUTCOMES:
Rates of abstinence of vaginal or anal sex | 3 months post intervention
  Reported number of times having had vaginal or anal intercourse. Response options range from 1 "Never" and 5 "4 or more times".
Rates of abstinence of vaginal or anal sex | 9 months post intervention
  Reported number of times having had vaginal or anal intercourse. Response options range from 1 "Never" to 5 "4 or more times".
Frequency of communicating without abuse | 3 months post intervention
  Reported number of times communicating with a partner without abuse. Response options range from 1 "Never - this has never happened in your relationship" to 4 "Often: this has happened 6 times or more in your relationship".
Frequency of communicating without abuse | 9 months post intervention
  Reported number of times communicating with a partner without abuse. Response options range from 1 "Never - this has never happened in your relationship" to 4 "Often: this has happened 6 times or more in your relationship".
Clinic utilization | 3 months post intervention
  Number of times receiving services or information from school-based health center on contraception, pregnancy, abortion, or sexually transmitted diseases
Clinic utilization | 9 months post intervention
  Number of times receiving services or information from school-based health center on contraception, pregnancy, abortion, or sexually transmitted diseases.
Behavioral intentions to engage in sexual activity | 3 months post intervention
  4 items from the Sexual Behavior Index (SBI) that assess one's willingness and intention to engage in sex in the next 3 months. Response options range from 1-7 with lower scores indicating lower willingness or intentions to engage in sexual activity.
Behavioral intentions to engage in sexual activity | 9 months post intervention
  4 items from the Sexual Behavior Index (SBI) that assess one's willingness and intention to engage in sex in the next 9 months. Response options range from 1-7 with lower scores indicating lower willingness or intentions to engage in sexual activity.
Behavioral intentions to use condoms | 3 months post intervention
  Assessed using 3 items from the COMPAS Program Behavioral Intentions Scale designed to measure one's intentions to acquire, discuss, and use condoms before sex. Items response options range from 1-4 with higher scores indicating higher intentions to perform the health behavior.
Behavioral intentions to use condoms | 9 months post intervention
  Assessed using 3 items from the COMPAS Program Behavioral Intentions Scale designed to measure one's intentions to acquire, discuss, and use condoms before sex. Items response options range from 1-4 with higher scores indicating higher intentions to perform the health behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Karin K Coyle, PhD, Principal Investigator — ETR; Pamela M Anderson, PhD, Principal Investigator — ETR
Locations (3):
- United States (3):
  - California School Based Health Alliance, Oakland, California
  - San Diego State University, San Diego, California
  - ETR, Scotts Valley, California

IPD SHARING:
Plan to Share IPD: No
As part of our commitment to data security and confidentiality, IPD will not be shared outside the research team.

REFERENCES:
- [Derived] Anderson P, Coyle K, Guinosso S, Ferrand JL, Owora A, Houghton RF, Walsh-Buhi E. Promoting Adolescent Healthy Relationships (The About Us Program): Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2021 Sep 1;10(9):e30499. doi: 10.2196/30499. PMID 34468330